CLINICAL TRIAL: NCT03044340
Title: Vascular and Neurologic Exploration of Small Nervous Fiber by Sudoscanner
Brief Title: Vascular and Neurologic Exploration of Small Nervous Fiber by Sudoscanner and QST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ERYTHROMELALGY
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Erythermalgia
MeSH Terms: conditions — Erythromelalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- erythermalgia patient (Experimental): patient will be measured chlorine ions impedance with the SUDOSCAN and evaluation on pain du to temperature with the THERMOTEST
  Interventions: Other: impedance measurement and pain evaluation

INTERVENTIONS:
Other: impedance measurement and pain evaluation — Measurement of chlorine ions impedance by SUDOSCAN and pain due to temperature evaluation with THERMOTEST

SUMMARY:
Erythromelalgy (EM) is a vascular syndrome very rare affecting the feet. This disease evolve by crisis when the feet extremities become red hot and painful. There are several types of EM but this study concern the adult primitive form. For a long time, the physiopathology was not described but now we know that there is a vascular form, with microcirculatory dysfunction and a neurologic form with small fibers neuropathy. The diagnostic of neurologic form is based on clinical evaluation (DN4 questionnaire, UENS scale...) and an electromyography. Thermotest, a medical device which measure the thermic sensitivity is used to quantify neuropathy. More recently Sudoscan, a device measuring cutaneous impedance to chloride ions detect small nervous fiber in diabetic patients with good correlation with Thermotest.

The purpose of this study is to analyze the vascular side and the neurologic side on patients consulting for Erythromelalgy.

ELIGIBILITY:
Inclusion Criteria:

* Pain with burn feeling at hands and feet extremities
* Crisis activated by the heat
* Age > 18 years old

Exclusion Criteria:

* Patients who had burn in extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Assessment of Chlorine ion production change | Day1
  patient will be measured the impedance of chlorinates ions by Sudoscan
Assessment of Temperature changing sensitivity | Day1
  Patients will be measured their sensitivity to temperature changing using the Thermotest

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No